Date of document: 11.16.17

## Study title:

1550-nm Non-Ablative Laser (Fraxel) Versus Ablative 10,600-nm Carbon Dioxide (CO<sub>2</sub>) Fractional Laser in the Treatment of Surgical and Traumatic Scars: A Comparison Study on Efficacy and Treatment Regimen.

NCT number: NCT02988622

